CLINICAL TRIAL: NCT05574998
Title: Recombinant Human Endostatin in Combination With Platinum-Based Doublet Chemotherapy for First-Line Treatment of Advanced Non-Small-Cell Lung Cancer With Negative Driver Gene: a Multicenter, Single-Arm Trial
Brief Title: First-Line Treatment of Advanced Non-Small-Cell Lung Cancer With Negative Driver Gene: a Multicenter, Single-Arm Trial
Acronym: FTANLCNDG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Degan Lu, professor, Qianfoshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2020(073); ChiCTR2100042088 (Registry Identifier: ChineseClinicalTrialRegistry)
Record Dates: First submitted 2022-10-06; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Non-Small-Cell Lung Cancer; Recombinant human endostatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Endostatins; endostar protein; Carboplatin; Cisplatin; Pemetrexed; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant Human Endostatin(Endostar) in Combination With Platinum-Based Doublet Chemotherapy (Experimental): The specific treatment regimen is as follows: Non-squamous NSCLC: Endostar (210 mg, CIV for 120 h) is started on the first day of each treatment cycle and administered every three weeks. Carboplatin AUC 5-6 mg/ml/min or cisplatin 75 mg/m2 (d4) +pemetrexed 500 mg/m2 (d4) Q3W is administered in this regimen for 4 cycles followed by Endostar plus pemetrexed until disease progression or intolerable toxicity.
  Squamous NSCLC: Endostar (210 mg, CIV for 120 hours) is started on the first day of each treatment cycle and administered every three weeks. Carboplatin AUC 5-6 mg/ml/min or cisplatin 75 mg/m2 (d4) + paclitaxel 175 mg/m2 (d4) Q3W.Endostar is administered after 4 cycles of this treatment regimen until disease progression or intolerable toxicity developed.
  Interventions: Drug: Recombinant human endostatin (Endostar)

INTERVENTIONS:
Drug: Recombinant human endostatin (Endostar) — The specific treatment regimen is as follows: Non-squamous NSCLC: Endostar (210 mg, CIV for 120 h) is started on the first day of each treatment cycle and administered every three weeks. Carboplatin AUC 5-6 mg/ml/min or cisplatin 75 mg/m2 (d4) +pemetrexed 500 mg/m2 (d4) Q3W is administered in this regimen for 4 cycles followed by Endostar plus pemetrexed until disease progression or intolerable toxicity.
  Squamous NSCLC: Endostar (210 mg, CIV for 120 hours) is started on the first day of each treatment cycle and administered every three weeks. Carboplatin AUC 5-6 mg/ml/min or cisplatin 75 mg/m2 (d4) + paclitaxel 175 mg/m2 (d4) Q3W.Endostar is administered after 4 cycles of this treatment regimen until disease progression or intolerable toxicity developed.
  Other Names: Carboplatin; Cisplatin; Pemetrexed; Paclitaxel

SUMMARY:
To evaluate the efficacy and safety of recombinant human endostatin (Endostar) combined with platinum-based doublet chemotherapy as the first-line therapy for patients with driver-gene-negative advanced non-small cell lung cancer(NSCLC).

This study is an exploratory single-arm study. The specific treatment regimen is as follows: Non-squamous NSCLC: Endostar (210 mg, continuous intravenous infusion (CIV) for 120 h) is started on the first day of each treatment cycle and administered every three weeks. Carboplatin AUC 5-6 mg/ml/min or cisplatin 75 mg/m2 (d4) +pemetrexed 500 mg/m2 (d4) Q3W is administered in this regimen for 4 cycles followed by Endostar plus pemetrexed until disease progression or intolerable toxicity.

Squamous NSCLC: Endostar (210 mg, continuous intravenous infusion (CIV) for 120 hours) is started on the first day of each treatment cycle and administered every three weeks. Carboplatin AUC 5-6 mg/ml/min or cisplatin 75 mg/m2 (d4) + paclitaxel 175 mg/m2 (d4) Q3W.Endostar is administered after 4 cycles of this treatment regimen until disease progression or intolerable toxicity developed.

Patients are assessed for measurable disease at baseline, 6 weeks, 12 weeks after starting treatment, and every 9 weeks thereafter according to RECIST 1.1 criteria during the treatment period until disease progression or intolerable toxicity withdrawal. Following discontinuation of treatment, subjects are followed for survival status every 3 months until death. Subject safety was assessed during treatment according to NCI CTCAE Version 4.0 criteria. Subjects who experience an AE should be followed until the AE returns to baseline. The primary endpoints is Progression-free survival (PFS) . Secondary endpoints include objective response rate (ORR), overall survival (OS) and safety (NCI CTCAE v 4.0).

Statistical methods: The PFS curve was estimated using the Kaplan-Meier method for the largest population to be analyzed. The confidence interval method was used as the criterion for the main analysis. OS was calculated in the same way as the secondary endpoint. Descriptive statistics will be used to analyze ORR, DCR, etc.

It is expected that continuous intravenous Endostar combined with platinum-based doublet chemotherapy as first-line treatment will prolong median PFS and OS in patients with driver gene-negative advanced NSCLC.

DETAILED DESCRIPTION:
With the progress of molecular biology and translational medicine research, the treatment of advanced non-small cell lung cancer(NSCLC) has entered the era of individualized treatment. EGFR-TKIs bring about 2 years of overall survival (OS) to patients with EGFR mutated advanced non-small cell lung cancer, and ALK mutations are also promising. For patients with lung cancer whose EGFR and ALK mutations are -negative or unknown, chemotherapy remains the mainstay of treatment. Platinum-based chemotherapy entered the plateau of efficacy.

The occurrence of tumor vessels depends on the activation, proliferation, adsorption and maturation process of vascular endothelial cells, all of which can be the target of vascular inhibitors. Recombinant human endostatin (Endostar) can inhibit tumor endothelial cell proliferation, angiogenesis and tumor growth. Endostar has been shown to be efficient and safe in the treatment of NSCLC and was approved by Chinese Food and Drug Administration. Endostar combined with platinum-based chemotherapy in non-small cell lung cancer has shown high safety and efficacy, with encouraging clinical application prospects. Endostar is currently administered in clinical application at 7.5 mg/m2 by instillation for 3 - 4 hours per day for 14 consecutive days as a cycle. Because its half-life is only about 10 hours, it will cause excessive fluctuations in plasma concentrations in the body and inability to maintain steady-state concentrations, while the patient 's compliance is also poor. Continuous intravenous infusion of Endostar can maintain steady-state plasma concentration and continuously inhibit tumor angiogenesis without increasing the toxicity of the drug, further improving the efficacy of Endostar and patient compliance. Although very low quality of evidence supported the survival benefit of continuous intravenous compared with intermittent intravenous, we need more evidence to demonstrate survival benefits.

Objective: To evaluate the efficacy and safety of Endostar(210 mg, continuous intravenous infusion(CIV) for 120h) combined with platinum-based doublet chemotherapy as the first-line therapy for patients with driver-gene-negative advanced NSCLC.

The research idea starts from the safety and efficacy of Endostar in vascular targeted therapy for lung cancer. Under the theoretical perspective of clinical research on cancer treatment, an exploratory multicenter single-arm study method is used to perform Endostar (210 mg, CIV 120h) combined with platinum-based chemotherapy regimen for first-line treatment of advanced NSCLC patients with negative driver gene. A database is established for the enrolled case report form, systematic data analysis is performed, and finally the study conclusions of Endostar safety, efficacy, timing method and optimization are obtained. It is expected that continuous intravenous Endostar combined with platinum-based doublet chemotherapy as first-line treatment will prolong median PFS and OS in patients with driver gene-negative advanced NSCLC.

This study is an exploratory single-arm study. The specific treatment regimen is as follows: Non-squamous NSCLC: Endostar (210 mg, CIV for 120 h) is started on the first day of each treatment cycle and administered every three weeks. Carboplatin AUC 5-6 mg/ml/min or cisplatin 75 mg/m2 (d4) +pemetrexed 500 mg/m2 (d4) Q3W is administered in this regimen for 4 cycles followed by Endostar plus pemetrexed until disease progression or intolerable toxicity.

Squamous NSCLC: Endostar (210 mg, CIV for 120 hours) is started on the first day of each treatment cycle and administered every three weeks. Carboplatin AUC 5-6 mg/ml/min or cisplatin 75 mg/m2 (d4) + paclitaxel 175 mg/m2 (d4) Q3W.Endostar is administered after 4 cycles of this treatment regimen until disease progression or intolerable toxicity developed.

Patients are assessed for measurable disease at baseline, 6 weeks, 12 weeks after starting treatment, and every 9 weeks thereafter according to RECIST 1.1 criteria during the treatment period until disease progression or intolerable toxicity withdrawal. Following discontinuation of treatment, subjects are followed for survival status every 3 months until death. Subject safety was assessed during treatment according to NCI CTCAE Version 4.0 criteria. Subjects who experience an AE should be followed until the AE returns to baseline.The primary endpoints is Progression-free survival (PFS) . Secondary endpoints include objective response rate (ORR), overall survival (OS) and safety (NCI CTCAE v 4.0).

Statistical methods: The PFS curve was estimated using the Kaplan-Meier method for the largest population to be analyzed. The confidence interval method was used as the criterion for the main analysis. OS was calculated in the same way as the secondary endpoint. Descriptive statistics will be used to analyze ORR, DCR, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic NSCLC is histologically or cytologically proven to be inoperable and cannot receive radical concurrent chemoradiotherapy. The conventional TNM stage was identified as stage IIIa-Ⅳb according to the International Association for the Study of Lung Cancer and the American Joint Committee on the Classification of Cancer 8th edition TNM Staging of Lung Cance.
2. The molecular testing for EGFR mutation,ALK and ROS1 is all negative.
3. Patients who had not previously received systemic radiotherapy and chemotherapy or who had relapsed for more than 6 months of follow-up after onset of adjuvant chemotherapy.
4. At least one measurable lesion as determined by RECIST criteria.
5. Male or female patients, age: 18-75 years of age.
6. Performance score 0-1 based on Eastern Cooperative Oncology Group (ECOG) test.
7. Expected survival period >= 12 weeks.
8. Serum absolute number of neutrophils >= 1.5 x 10^9/L, platelet >= 100 x 10^9/L,and hemoglobin >= 90g/L.
9. Serum bilirubin <= 1.5 times ULNL, aspartate aminotransferase (AST) and adenosine triphosphate(ALT) <= 2.5 times ULN, alkaline phosphatase <= 5 times ULN.
10. Serum creatinine <= the ULN or creatinine clearance >= 60 mL/min.
11. Patients who had previously undergone surgery have recovered for more than 4 weeks from the beginning of the project.
12. Women with an intact uterus must have a negative pregnancy test within 28 days prior to enrolement in the study (unless it was 24 months after amenorrhea). If the pregnancy test is more than 7 days prior to initial dosing, a urine pregnancy test is required for verification (within 7 days prior to initial dosing).
13. Sign the inform consent form with good compliance. Exclusion criteria：

1.Intolerance to platinum therapy or allergy to platinum drugs. 2.Allergic to recombinant human endostatin (endostar) and its any components. 3.Pregnancy or breastfeeding women or women who may be pregnant but are unwilling to take appropriate contraception.

4.Existing severe acute infections that are not under control; Or suppurative and chronic infections with delayed healing.

5.Pre-existing serious heart disease, including: congestive heart failure, uncontrolled high-risk arrhythmias, unstable angina pectoris, myocardial infarction, severe valvular heart disease, and refractory hypertension.

6.People suffering from uncontrollable neuropsychiatric diseases or mental disorders had poor compliance and were unable to cooperate and describe treatment responses; The conditions of patients with primary brain tumor or central nerve metastatic tumor were uncontrollable and the symptoms of cranial hypertension or neuropsychiatric were obvious.

7.People with tendency of bleeding. 8.Other conditions that the investigator considers to be inappropriate for the patient to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  Progression-free survival

SECONDARY OUTCOMES:
OS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  overall survival
ORR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Degan Lu, professor, Principal Investigator — Shandong First Medical University
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Result] Rinaldi M, Cauchi C, Gridelli C. First line chemotherapy in advanced or metastatic NSCLC. Ann Oncol. 2006 May;17 Suppl 5:v64-7. doi: 10.1093/annonc/mdj953. PMID 16807466
- [Result] Wang J, Sun Y, Liu Y, Yu Q, Zhang Y, Li K, Zhu Y, Zhou Q, Hou M, Guan Z, Li W, Zhuang W, Wang D, Liang H, Qin F, Lu H, Liu X, Sun H, Zhang Y, Wang J, Luo S, Yang R, Tu Y, Wang X, Song S, Zhou J, You L, Wang J, Yao C. [Results of randomized, multicenter, double-blind phase III trial of rh-endostatin (YH-16) in treatment of advanced non-small cell lung cancer patients]. Zhongguo Fei Ai Za Zhi. 2005 Aug 20;8(4):283-90. doi: 10.3779/j.issn.1009-3419.2005.04.07. Chinese. PMID 21108883
- [Result] Zhai Y, Ma H, Hui Z, Zhao L, Li D, Liang J, Wang X, Xu L, Chen B, Tang Y, Wu R, Xu Y, Pang Q, Chen M, Wang L. HELPER study: A phase II trial of continuous infusion of endostar combined with concurrent etoposide plus cisplatin and radiotherapy for treatment of unresectable stage III non-small-cell lung cancer. Radiother Oncol. 2019 Feb;131:27-34. doi: 10.1016/j.radonc.2018.10.032. Epub 2018 Dec 17. PMID 30773184
- [Result] Hansma AH, Broxterman HJ, van der Horst I, Yuana Y, Boven E, Giaccone G, Pinedo HM, Hoekman K. Recombinant human endostatin administered as a 28-day continuous intravenous infusion, followed by daily subcutaneous injections: a phase I and pharmacokinetic study in patients with advanced cancer. Ann Oncol. 2005 Oct;16(10):1695-701. doi: 10.1093/annonc/mdi318. Epub 2005 Jul 12. PMID 16012180
- [Derived] Liu X, Guo Z, Su L, Zuo A, Gao M, Ji X, Lu J, Yang S, Jiang Y, Lu D. The efficacy and safety of continuous intravenous infusion of rh-endostatin combined with platinum-based doublet chemotherapy for advanced non-small-cell lung cancer. Invest New Drugs. 2024 Jun;42(3):309-317. doi: 10.1007/s10637-024-01439-x. Epub 2024 May 3. PMID 38700579
- See also: N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. — https://pubmed.ncbi.nlm.nih.gov/19692680/
- See also: Ann Oncol. 2006 May;17 Suppl 5:v64-7. Review. — https://pm.yuntsg.com/searchList.html
- See also: Zhongguo Fei Ai Za Zhi. 2005 Aug 20;8(4):283-90. — https://pm.yuntsg.com/searchList.html
- See also: Radiother Oncol. 2019 Feb;131:27-34 — https://pubmed.ncbi.nlm.nih.gov/30773184/
- See also: Ann Oncol. 2005 Oct;16(10):1695-701. Epub 2005 Jul 12. — https://pm.yuntsg.com/searchList.html